CLINICAL TRIAL: NCT07079956
Title: A Prospective, Single-Arm, Multicenter, Feasibility Trial to Evaluate the Safety and Performance of the TUBE Device in the Endovascular Treatment of Unruptured, Wide-Neck or Fusiform Intracranial Aneurysms
Brief Title: Study to Evaluate the TUBE Device Ability to Treat Unruptured, Wide-neck or Fusiform Aneurysms
Acronym: NV01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NVMedTech (Industry)
Collaborators: BioMDg (Unknown); RARAS CRO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV01
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Aneurysm Cerebral
Keywords: Aneurysm; Wide-neck; Fusiform; Flow Diverter
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Masking Description: Clinical Events Committee (CEC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Eligible participants will receive treatment with the TUBE Flow Diverter device (Experimental): the TUBE device is for the treatment of unruptured, saccular wide-neck or fusiform intracranial aneurysms arising from a parent vessel with a diameter ≥ 2.0 mm and ≤ 5.0 mm and located on the ICA or its branches.
  Interventions: Device: TUBE Flow Diverter

INTERVENTIONS:
Device: TUBE Flow Diverter — TUBE Device

SUMMARY:
To assess the safety and performance of the TUBE device in the endovascular treatment of unruptured, wide-neck or fusiform intracranial aneurysms located on the internal carotid artery (ICA) or its branches

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter study designed to assess the safety and performance of the TUBE device in the endovascular treatment of unruptured, saccular wide-neck (neck width ≥ 4 mm or dome-to-neck ratio < 2) or fusiform intracranial aneurysms arising from a parent vessel with a diameter ≥ 2.0 mm and ≤ 5.0 mm and located on the ICA or its branches.

Up to 20 eligible patients who present for flow diverter placement, provide informed consent, meet all inclusion crite-ria, and not meet any exclusion criteria will receive treatment with the TUBE device. All participants will be followed for 1 year. Post-procedure, imaging will be repeated at the Day 30, Month 3, 6, and 12 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Has a single unruptured target intracranial aneurysm (IA) with the following characteristics:

   1. Is located on the internal carotid artery or its branch-es.
   2. Has a neck ≥ 4 mm, dome to neck ratio < 2.0, or no discernible neck
   3. Aneurysm diameter ≤ 35 mm (saccular or fusiform configuration)
2. Has a parent vessel diameter ≥ 2.0 mm and ≤ 5.0 mm at both the proximal and distal segments where the implant will be placed.
3. Has multiple increased risk factors for intracranial aneurysm rupture, including but not limited to, aneurysm morphology, smoking, hypertension, diabetes, age, prior and/or family history of aneurysm rupture, and/or history of subarachnoid hemorrhage that may result in a benefit risk profile of endovascular treatment that outweighs the risks of intracranial aneurysm rupture during the patient's expected lifetime if left untreated.
4. The patient is able and willing to provide written in-formed consent.

Exclusion Criteria:

Participants are not eligible for the study if ANY of the following criteria are present:

1. Has an extradural aneurysm
2. Has a target aneurysm in the posterior circulation
3. Perforator or branch vessel, inclusive of the posterior communicating artery, arises from the target aneurysm body or neck (branches or arteries must arise or connect from the parent vessel separate from the aneurysm or neck to not be excluded from study)
4. Has a true bifurcation aneurysm, defined as an aneurysm (saccular or non-saccular) located at a point of vessel bifurcation
5. Target aneurysm is unsuitable for flow diverter treatment
6. Has vessel characteristics, such as severe tortuosity (cICA Type IV), stenosis (>70%), or morphology that would preclude safe endovascular access to the target aneurysm necessary for treatment with the study device
7. Received previous treatment of the target aneurysm or parent artery where it would interfere with the placement or proper apposition of the device
8. Has a medical contraindication to study or procedure related antiplatelet medications (aspirin, clopidogrel/ Plavix, prasugrel, ticagrelor, and heparin), local or general anesthesia, or life-threatening allergy to contrast dye
9. Non-responders to prasugrel as determined by the P2Y12 assay ("VerifyNow" system)
10. Has a known severe allergy to nickel titanium, stainless steel (304SS) tantalum, or platinum.
11. Modified Rankin Score assessment is ≥ 3 at pre-procedure exam
12. Presence of unstable neurological deficit (i.e., worsening of clinical condition in the last 30 days)
13. Subarachnoid hemorrhage occurred within 30 days prior to enrollment
14. Major surgery (including previous intracranial implant) occurred within previous 30 days or is planned in the next 120 days after enrollment date
15. Has more than one intracranial aneurysm that requires treatment within 12 months
16. Received previous intracranial implant associated with the symptomatic or vascular distribution within the past 12 weeks prior to treatment date
17. Chronic anticoagulation therapy is ongoing or known coagulopathy exists
18. Has other known serious concurrent medical conditions such as heart disease (e.g., atrial fibrillation [with or without pacemaker], recent myocardial infarction [< 12 weeks ago], symptomatic congestive heart failure, or carotid stenosis), kidney failure [>2.0mg/dl serum creatinine], pulmonary disease, uncontrolled diabetes, progressive neurologic disorders, terminal cancer, vasculitis, high risk of ischemic stroke or recent stroke
19. Has acute life-threatening illness other than the neurological disease (e.g., acute kidney or heart failure) to be treated in this trial
20. Life expectancy is less than 5 years due to other illness or condition (in addition to an intracranial aneurysm)
21. Unable to complete study follow up due to dementia or psychiatric problem, substance abuse, or history of noncompliance with medical advice
22. Pregnancy at time of enrollment
23. Presence of intracranial mass (tumor, except meningioma, abscess, or other infection), non-treated arteriovenous malformation (AVM) in the territory of the target aneurysm
24. Evidence of active infection at the time of treatment
25. Enrollment in another trial involving an investigational product that could confound the outcomes of this trial.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Neurologic death, or disabling stroke | At 12 months
  Primary Safety Outcome
Primary Performance Outcome | At 12 months post-procedure
  The proportion of participants with composite of 100% occlusion (Raymond-Roy Classification 1, complete occlusion) of the target aneurysm without significant parent artery stenosis (> 50% stenosis) on digital subtraction angiography (DSA) images.

SECONDARY OUTCOMES:
Performance Outcome | 1 month, 3 months, and 6 months post-procedure respectively
  The proportion of participants with composite of 100% occlusion (Raymond-Roy Classification 1, complete occlusion) of the target aneurysm without significant parent artery stenosis (> 50% stenosis) and with no retreatment of the target aneurysm.

CONTACTS AND LOCATIONS:
Overall Officials: Michel E. Frudit, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina da USP
Locations (3):
- Brazil (3):
  - Hospital Geral de Fortaleza, Fortaleza
  - Instituto Estadual do Cérebro Paulo Niemeyer, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo

IPD SHARING:
Plan to Share IPD: No